CLINICAL TRIAL: NCT00765596
Title: Ghrelin Changes After Roux-en-Y Gastric Bypass: Does Gastric Pouch vs. Gastric Remnant Feeding Affect Secretion?
Brief Title: Ghrelin Changes After Roux-en-Y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Naji Abumrad, Chairman, Department of Surgery, Vanderbilt University
Other Study IDs: IRB#041129
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Insulin resistance; Gastric tube; Ghrelin
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 RYGB: Subjects undergoing RYGB with gastric tube placement
- 2 Matched controls: Subjects matched by BMI, age, gender to RYGB group
  Interventions: Other: Liquid diet for 3 days

INTERVENTIONS:
Other: Liquid diet for 3 days — The control group were given a 3 -day liquid diet similar to the RYGB post-op diet
  Groups: 2 Matched controls

SUMMARY:
The purpose of this study is to determine whether gastric division (via Roux-en-Y gastric bypass) with resultant fundic isolation will alter the pattern(s) of Ghrelin secretion in the early post-operative period following feeding in morbidly obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine and liver function tests < upper limits of normal
* Stable body weights for the past three months
* Women will have a negative pregnancy test
* patients who are already scheduled for RYGB with gastrostomy tube placement

Exclusion Criteria:

* Significant hepatic enzyme elevations (more than 100% of upper limits of normal)
* Serum creatinine > 1.5 mg/dl
* history of ketoacidosis or current metabolic acidosis
* current use of oral anticoagulants
* Positive pregnancy test (beta-human chorionic gonadotrophin) for females
* intercurrent infections
* patients with prior gastric operations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects were morbidly obese, scheduled for RYGB with gastric tube placement. Controls were matched to subjects by BMI, age, gender.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Ghrelin | pre-op, peri-op, immediately post-op, 2 days, 3 wks, 6wks, 6mos, 1 year post op

SECONDARY OUTCOMES:
HOMA | pre-op, peri-op, immediately post-op, 2 days, 3 wks, 6wks, 6mos, 1 year post op
metabolic hormones | pre-op, peri-op, immediately post-op, 2 days, 3 wks, 6wks, 6mos, 1 year post op

CONTACTS AND LOCATIONS:
Overall Officials: Naji N Abumrad, MD, Principal Investigator — Department of Surgery, Vanderbilt University Medical Center; Erik N Hansen, MD, Principal Investigator — Departement of Surgery, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Hansen EN, Tamboli RA, Isbell JM, Saliba J, Dunn JP, Marks-Shulman PA, Abumrad NN. Role of the foregut in the early improvement in glucose tolerance and insulin sensitivity following Roux-en-Y gastric bypass surgery. Am J Physiol Gastrointest Liver Physiol. 2011 May;300(5):G795-802. doi: 10.1152/ajpgi.00019.2011. Epub 2011 Mar 3. PMID 21372167
- [Derived] Isbell JM, Tamboli RA, Hansen EN, Saliba J, Dunn JP, Phillips SE, Marks-Shulman PA, Abumrad NN. The importance of caloric restriction in the early improvements in insulin sensitivity after Roux-en-Y gastric bypass surgery. Diabetes Care. 2010 Jul;33(7):1438-42. doi: 10.2337/dc09-2107. Epub 2010 Apr 5. PMID 20368410